CLINICAL TRIAL: NCT06788769
Title: Retrospective Analysis of Risk Factors and Microbiome Alterations in Infant Clostridioides Difficile Infection
Brief Title: Study of Clostridioides Difficile in Infants
Status: Recruiting | Type: Observational
Sponsor: Westlake University (Other)
Responsible Party: Sponsor
Other Study IDs: 20241202TL001
Record Dates: First submitted 2025-01-16; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Clostridioides Difficile Infection
Keywords: Clostridioides Difficile; Infants
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (3):
- CDI Patients: This group includes infants aged 0-2 years who have been diagnosed with Clostridioides difficile infection (CDI). Diagnosis is based on clinical symptoms such as diarrhea, abdominal pain, or fever, along with positive laboratory confirmation (e.g., stool PCR or culture for C. difficile).
- Asymptomatic Clostridioides difficile Carriers: This group includes infants aged 0-2 years who are colonized with Clostridioides difficile but show no clinical symptoms of infection. Participants in this group tested positive for C. difficile in fecal samples collected during routine or study-related screening.
- Healthy Infants: This group includes infants aged 0-2 years who do not show any clinical symptoms of infection and have tested negative for Clostridioides difficile in fecal samples. Participants were recruited from general pediatric clinics or community health programs.

SUMMARY:
Clostridioides difficile infection (CDI) poses an increasing threat to infant and young child health, with detection rates rising annually. This retrospective study aims to explore the epidemiological characteristics, clinical manifestations, and potential biomarkers of CDI in children aged 0-2 years by examining three cohorts: (1) infants diagnosed with CDI, (2) asymptomatic carriers of C. difficile, and (3) healthy controls. Fecal samples from each group will undergo metagenomic sequencing and metabolomic profiling, coupled with questionnaire-based surveys for risk factor assessment. The findings are anticipated to identify key high-risk factors, elucidate the pathogenic mechanisms underlying infant CDI, and support the development of early diagnostic tools and preventive strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Age Range: Infants aged 0 to 2 years (inclusive) at the time of sample collection or medical record documentation.
2. Data Availability: Complete medical records or available stool samples within the study's retrospective time frame.
3. Group-Specific Criteria:

   CDI Patients: Documented diarrhea or related gastrointestinal symptoms, with laboratory-confirmed C. difficile by PCR or culture.

   Asymptomatic Carriers: Positive C. difficile test (PCR or culture) in the absence of diarrhea or other clinical CDI symptoms.

   Healthy Controls: Negative C. difficile test and no gastrointestinal symptoms indicative of CDI.
4. Consent/Authorization:Retrospective data (e.g., existing medical records or stored biosamples) may be included under a waiver of consent if approved by the institutional review board (IRB). However, any new information obtained directly from participants or their guardians (e.g., via questionnaires) requires explicit informed consent.

Exclusion Criteria:

1. Incomplete Data: Infants whose medical records lack sufficient information to confirm their CDI status or those without adequate stool sample results.
2. Ambiguous Diagnosis: Patients presenting with other infectious diseases or conditions that could not rule out alternative diagnoses for diarrhea (e.g., confirmed concurrent viral or parasitic infections) without conclusive C. difficile testing.
3. Severe Comorbidities: Infants with life-threatening congenital conditions (e.g., severe immunodeficiency syndromes) if these conditions significantly alter the gut microbiota or confound CDI diagnosis.

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This retrospective observational study will include infants aged 0 to 2 years who underwent clinical evaluation and stool testing for Clostridioides difficile at [Hospital(s)/Institution(s)/Region]. The study population is divided into three groups:
  1. CDI Patients: Infants with laboratory-confirmed C. difficile (PCR or culture) and clinical symptoms consistent with infection (e.g., diarrhea, abdominal pain).
  2. Asymptomatic Carriers: Infants who tested positive for C. difficile but did not exhibit any related symptoms.
  3. Healthy Controls: Infants who tested negative for C. difficile and had no history of gastrointestinal symptoms during the same period.
  All participants included in this analysis will have relevant medical records and stool sample data available within the study's retrospective timeframe. Additional questionnaire data may be collected from parents or guardians to assess potential risk factors and environmental exposures
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Clostridioides difficile infection (CDI) and asymptomatic carriage in infants | Data from medical records and stool sample tests collected retrospectively between July 2024 and December 2026.
  The prevalence of CDI and asymptomatic C. difficile carriage will be determined by testing fecal samples for C. difficile using PCR and/or culture methods. Participants are categorized into three groups based on clinical symptoms (diarrhea, abdominal pain, or fever) and laboratory confirmation (positive PCR or stool culture).
  Specifically, the primary outcome assesses:
  1. The proportion of infants (0-2 years) testing positive for C. difficile who exhibit clinical symptoms (CDI patients).
  2. The proportion of infants (0-2 years) testing positive but showing no symptoms (asymptomatic carriers), and the proportion of infants testing negative (healthy controls).

SECONDARY OUTCOMES:
Gut Microbial Diversity Among CDI Patients, Asymptomatic Carriers, and Healthy Controls | Same retrospective collection period (2024-2026)
  Metagenomic sequencing will be performed on fecal samples to assess alpha and beta diversity.The goal is to compare microbial community shifts and identify specific taxa changes associated with CDI.

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No